CLINICAL TRIAL: NCT02896738
Title: MRI Screening for Auditory Pathway Malformations in Visually Impaired Children
Acronym: DIMAVE
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: LBU_2015_6
Record Dates: First submitted 2016-09-07; First posted 2016-09-12 (Estimated); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Visual Impairment
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
This pilot study aims to assess the interest to add an auditory pathway morphological analysis during the MRI exploration of visual pathway in visually impaired children.

ELIGIBILITY:
Inclusion Criteria:

* age < 18 years old
* visual impairment
* MRI scheduled to explore their visual impairment
* parents' informed consent for participation in the study

Exclusion Criteria:

* tumoral origin for the visual impairment
* no health insurance coverage

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Visually impaired children undergoing MRI exploration.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-04-12 (Actual)

PRIMARY OUTCOMES:
number of patients with Auditory Pathway Malformation | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Louise Boyeldieu, MD, Principal Investigator — Fondation OPH A de Rothschild
Locations (1):
- Fondation Ophtalmologique Adolphe de Rothschild, Paris, France